CLINICAL TRIAL: NCT04450589
Title: Hair Regrowth Efficacy of Multi-Molecular Targeting Treatment (ALRV5XR), a Randomized Controlled Clinical Trial in Men With Androgenetic Alopecia, Telogen Effluvium or Self Reported Thinning Hair: THE HAIR REBOOT TRIAL - MEN
Brief Title: A Study Evaluating the Hair Regrowth Efficacy and Safety of ALRV5XR in Male Subjects With Hair Loss
Acronym: REBOOT-MEN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Arbor Life Labs (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ALL-180001-01
Record Dates: First submitted 2020-06-25; First posted 2020-06-29 (Actual); Last update posted 2020-06-30 (Actual); Status verified 2020-06

CONDITIONS: Androgenetic Alopecia; Androgenic Alopecia; Telogen Effluvium; Thinning Hair; Hair Loss/Baldness; Hair Thinning
Keywords: Androgenetic Alopecia; Androgenic Alopecia; Alopecia; Androgenetic; Androgenic; Telogen; Telogen Effluvium; Hair Loss; Baldness; Male Patterned Balding; Aging; Ageing; Senescence; Wnt; Wnt Beta-catenin Signaling Pathway; Stem Cell
MeSH Terms: conditions — Alopecia

STUDY DESIGN:
Intervention Model Description: Subjects will be randomized into 1 of 2 parallel groups. There will be one (1) treatment group and one (1) placebo group. Subjects will receive either the ALRV5XR treatment regimen or placebo regimen.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Study agents will have randomized codes. Supplement capsules, shampoo, conditioner and scalp serum will all be similar in look and scent to the active products. The placebo shampoo, conditioner and serum will have the same base materials as their counterparts but will not contain active ingredients, and will therefore be similar in viscosity and color.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ALRV5XR (Active Comparator): The ALRV5XR (active) group will receive ALRV5XR active treatment. Study agents will have randomized codes. Supplement capsules, shampoo, conditioner and scalp serum will all be similar in look and scent to the placebo products.
  Interventions: Dietary Supplement: ALRV5XR; Other: ALRV5XR Shampoo; Other: ALRV5XR Conditioner; Other: ALRV5XR Hair Follicle Serum (Nutriment)
- Placebo (Placebo Comparator): The Placebo group will receive a placebo (vehicle) treatment. Study agents will have randomized codes. Supplement capsules, shampoo, conditioner and scalp serum will all be similar in look and scent to the active products. The placebo shampoo, conditioner and serum will have the same base materials (vehicle) as their counterparts but will not contain active ingredients, and will therefore be similar in viscosity and color.
  Interventions: Dietary Supplement: Placebo; Other: Placebo Shampoo; Other: Placebo Conditioner; Other: Placebo Hair Follicle Serum (Nutriment)

INTERVENTIONS:
Dietary Supplement: ALRV5XR — ALRV5XR oral supplement. Dose/Route/Schedule: 1 capsule/oral twice daily. Take one capsule in the morning and one capsule in the evening. Take 30-60 minutes before food. If stomach upset occurs, subjects will be instructed to take the capsule at the beginning of a meal.
  There should be no deviation from the daily nutriment regimen (although in the event a capsule or day is missed, subject should continue with regimen the following day.)
  Other Names: Replenology; Replenology Hair; 21 To Grow; Nutrient Replenishment Biology; Replenology Hair Professional; Replenology Professional; Replenology Restore
  Arms: ALRV5XR
Other: ALRV5XR Shampoo — ALRV5XR Shampoo. Dose/Route/Schedule: 3-7 ml, topical, daily. The amount of shampoo used will vary by subject, based on length of hair. Short hair will use approximately 3ml of shampoo per wash and long hair as much as 7 ml. For short hair, an amount equivalent to a quarter in the palm of a hand, and for long hair a half-dollar size.
  There should be no deviation from the daily nutriment regimen (although in the event a day is missed, subject should continue with regimen the following day
  Other Names: Replenology; Replenology Hair; Replenology Shampoo; Nutrient Replenishment Biology; 21 To Grow; Replenology Retain
  Arms: ALRV5XR
Other: ALRV5XR Conditioner — ALRV5XR Conditioner. Dose/Route/Schedule: 3-7 ml, topical, daily. The amount of conditioner used will vary by subject based on length of hair. Short hair will use approximately 3ml of conditioner per wash and long hair as much as 7 ml. For short hair, an amount equivalent to a quarter in the palm of a hand, and for long hair a half-dollar size.
  There should be no deviation from the daily nutriment regimen (although in the event a day is missed, subject should continue with regimen the following day
  Other Names: Replenology; Replenology Hair; Replenology Conditioner; Nutrient Replenishment Biology; 21 To Grow; Replenology Reinforce
  Arms: ALRV5XR
Other: ALRV5XR Hair Follicle Serum (Nutriment) — ALRV5XR topical Hair Follicle serum (Nutriment), sealed in an airless pump dispensing bottle, metered at 0.2ml per depression. Dose/Route/Schedule: 1ml, topical, daily, applied at night.
  Topical serum (referred to as the Nutriment) dosage is metered as 5 x depressions of plunger per day to cover areas of thinning scalp and adjacent scalp areas. Care should be taken to limit the Nutriment in hair. Each depression is metered at 0.2ml for a daily dose of 1.0 ml. Each container has 30ml of Nutriment. Nutriment will dry within a few minutes and any on the hair will also dry. The dried effect in the hair should not cause oiliness or dryness on scalp or hair. There should be no deviation from the daily nutriment regimen (although in the event a day is missed, subject should continue with regimen the following day.)
  Other Names: Replenology; Replenology Follicle Nutriment; Replenology Hair; Nutrient Replenishment Biology; 21 To Grow; Replenology Revitalize; Replenology Scalp Serum
  Arms: ALRV5XR
Dietary Supplement: Placebo — Placebo oral supplement. Dose/Route/Schedule: 1 capsule/oral twice daily. Take one capsule in the morning and one capsule in the evening. Take 30-60 minutes before food. If stomach upset occurs, subjects will be instructed to take the capsule at the beginning of a meal.
  There should be no deviation from the daily nutriment regimen (although in the event a capsule or day is missed, subject should continue with regimen the following day.)
  Arms: Placebo
Other: Placebo Shampoo — Placebo Shampoo. Dose/Route/Schedule: 3-7 ml, topical, daily. The amount of shampoo used will vary by subject, based on length of hair. Short hair will use approximately 3ml of shampoo per wash and long hair as much as 7 ml. For short hair, an amount equivalent to a quarter in the palm of a hand, and for long hair a half-dollar size.
  There should be no deviation from the daily nutriment regimen (although in the event a day is missed, subject should continue with regimen the following day
  Arms: Placebo
Other: Placebo Conditioner — Placebo Conditioner. Dose/Route/Schedule: 3-7 ml, topical, daily. The amount of conditioner used will vary by subject based on length of hair. Short hair will use approximately 3ml of conditioner per wash and long hair as much as 7 ml. For short hair, an amount equivalent to a quarter in the palm of a hand, and for long hair a half-dollar size.
  There should be no deviation from the daily nutriment regimen (although in the event a day is missed, subject should continue with regimen the following day
  Arms: Placebo
Other: Placebo Hair Follicle Serum (Nutriment) — Placebo topical Hair Follicle serum (Nutriment), sealed in an airless pump dispensing bottle, metered at 0.2ml per depression. Dose/Route/Schedule: 1ml, topical, daily, applied at night.
  Topical serum (referred to as the Nutriment) dosage is metered as 5 x depressions of plunger per day to cover areas of thinning scalp and adjacent scalp areas. Care should be taken to limit the Nutriment in hair. Each depression is metered at 0.2ml for a daily dose of 1.0 ml. Each container has 30ml of Nutriment. Nutriment will dry within a few minutes and any on the hair will also dry. The dried effect in the hair should not cause oiliness or dryness on scalp or hair. There should be no deviation from the daily nutriment regimen (although in the event a day is missed, subject should continue with regimen the following day.)
  Arms: Placebo

SUMMARY:
To demonstrate that the ALRV5XR multi-molecular targeting treatment regimen of a daily shampoo, conditioner, topical serum and oral supplement is superior to placebo in promoting hair growth as assessed by change in hair density and percentage of terminal hair regrowth after ALRV5XR therapy.

This will be a single-centre, double-blind, randomized, placebo-controlled study in male subjects randomized to a 1:1 ratio of test article to placebo.

Subjects will be asked to use the study products on a daily basis for the duration of the 24-week study. Subjects will take one capsule twice daily (one in the morning and one in the evening) and will be asked to use 3-7mL of the shampoo, 3-7mL of the conditioner, and 1mL of the topical nutriment daily. Subjects will receive detailed instructions regarding the order and duration of application of each product.

Subjects in the active arm will receive active capsules, shampoo, conditioner and topical nutriment. Subjects on placebo will receive placebo capsules, shampoo, conditioner and topical nutriment. All subjects will be instructed to take the capsules orally, one in the morning and one in the evening, prior to consuming food. Shampoo and conditioner are to be used once per day when washing the hair and nutriment applied at the end of the day prior to bedtime. To facilitate this, subjects will receive a 3-month supply of each product (supplement, shampoo, conditioner, and scalp nutriment). Subjects will continue the daily regimen for 24 weeks, visiting the clinic at week 12 for an interim assessment.

DETAILED DESCRIPTION:
This is a prospective, randomized, double-blind, placebo-controlled, 2-arm parallel study to evaluate the efficacy and safety of a multi-molecular targeting botanical treatment regimen on parameters of hair growth, compared to placebo, in healthy male adults with androgenetic alopecia, diffuse hair loss or self-reported thinning hair.

Each study group will include 23 subjects. Subjects will be randomly assigned using computer generated randomization scheme to one of the two groups in a 1:1 ratio.

Subjects will be asked to use the study products on a daily basis for the duration of the 24-week study. Subjects will take one capsule twice daily (one in the morning and one in the evening) and will be instructed to use 3-7mL of the shampoo, 3-7mL of the conditioner, and 1mL of the topical nutriment serum daily. Subjects will receive detailed instructions regarding the order, and duration of application of each product.

This trial will be conducted at one (1) American (USA) clinical research site. The duration of the study will be approximately 28 weeks (7 months), including the screening period. There will be a screening period of up to 28 days for eligibility assessment, followed by a baseline visit followed by a 24-week experimentation period for assessment of supplement effects. There will be a total of seven visits, including a screening visit, over this 28-week period.

The study will be conducted as outlined in this protocol and in compliance with the principles of the International Conference on Harmonization (ICH) Guidelines on Good Clinical Practice (GCP) (E.6), and the Declaration of Helsinki.

Prior to initiating any study-related procedures, each subject must provide written informed consent in accordance with Institutional Research Board (IRB) requirements and applicable regulations. Any potential subject will be contacted by a designated member of the research team at the study site. Potential subjects may complete a web-based pre-screening questionnaire or may be interviewed. During the interview (or web-based questionnaire), subjects will answer specific questions, in order to assess their eligibility. If they meet pre-screening requirements, they will be invited to schedule a screening visit (Visit 1) with a Study Coordinator no more than 30 days prior to the anticipated baseline visit (Visit 2). In the event that subjects' screening period exceeds 30 days, the Investigator may repeat blood work, biometrics and/or vital signs (as appropriate) to ensure that subjects remain eligible.

Visit 1 (Screening Visit):

At the screening visit (Visit 1), up to 30 days prior to the Baseline Visit (Visit 2), the overall details of the study and the procedures to be undertaken will be explained to the subject. The following information will be recorded and procedures carried out:

* Subject registration
* Informed Consent (copy to subject)
* Subject education/comprehension questionnaire
* Review inclusion & exclusion criteria
* Assess Fitzpatrick phototype skin classification
* Demographic data (dietary habits, race, ethnicity, age, etc.)
* Medical history
* Concomitant medications recorded
* Measure screening anthropometrics and vital signs: height (cm), weight (kg), temperature (°C) respiratory rate (breaths/min), blood pressure (mmHg) and heart rate (bpm).
* Calculate BMI (kg/m2)
* Scalp examination (including photographs) for each subject will include a screen for immediately observable medical issues and any scalp alopecia/scalp disorders; photography of hair (top, right side, left side, back) - photographs will be shared with the Sponsor for determination of eligibility to participate in the study.
* Physical examination (excluding breast, genital and anorectal exam)
* Collect fasting (>6h, nothing to eat or drink except water) blood for screening laboratory tests
* Provide the subject with an instruction handout explaining visit preparation and overall study requirements (provide written and verbal instructions).

Remind subjects to follow inclusion/exclusion criteria of restrictions for both OTC and prescription medications, maintain current dietary habits, sleep habits, exercise and sexual intercourse habits.

If the subject is eligible for the study, they will be given a date to attend the Site no more than 30 days after the screening visit.

Visit 2 (Baseline Visit) - Day 0 Inclusion/Exclusion Criteria will be re-assessed to ensure eligibility. Concomitant medications and adverse events (AE's) will be reviewed. Eligible subjects will be randomized to one of the two treatment arms.

The following procedures will be completed prior to dosing:

* Monitor adverse events (since the previous visit)
* Review concomitant medications
* Measure anthropometrics and vital signs: weight (kg), temperature (°C) respiratory rate (breaths/min), blood pressure (mmHg) and heart rate (bpm)
* Calculate BMI (kg/m2)
* Review inclusion & exclusion criteria
* Scalp examination (including photographs) for each subject will include a screen for observable medical issues and any skin/scalp disorders; photography of hair (top, right side, left side, back) - photographs will be reviewed and SALT score determined by a dermatologist. General photographic instructions are described in APPENDIX III.
* Subjects will be asked to complete the Dermatology Quality of Life Index (DQLI)
* Use Trichology device to capture images of scalp target area for efficacy assessments
* Randomize eligible subjects
* Provide subject with the first dose of the oral supplement in clinic

The following procedures will be completed after dosing:

* Monitor subject for any immediate reactions (minimum 15-minute observation post- administration)
* Dispense 3-month supply of investigational product
* Provide subjects with instruction for using kit contents
* Remind subjects to follow inclusion/exclusion criteria for restrictions for both OTC and prescription medications, maintain current dietary habits, sleep habits, exercise and sexual intercourse habits.
* Provide subjects with a diary to record product use and any changes to health status or medication use

Visit 3 (Return for anagen/telogen ratio assessment) - day 3 Subjects will return to the clinic on day 3 to have the baseline anagen/telogen ratio assessed.

Visit 4 (Interim Visit) - Day 84 Study subjects will return to the Clinic on Day 84.

The following procedures will be completed:

* Collect daily diaries and review
* Collected investigational product containers (used and unused) and assess compliance
* Monitor adverse events (since the previous visit)
* Review concomitant medications (including changes to medications, changes to dose and frequency)
* Measure anthropometrics and vital signs: weight (kg), temperature (°C) respiratory rate (breaths/min), blood pressure (mmHg) and heart rate (bpm)
* Calculate BMI (kg/m2)
* Scalp examination (including photographs) for each subject will include a screen for observable medical issues and any skin/scalp disorders; photography of hair (top, right side, left side, back) - photographs will be reviewed and SALT score determined by a dermatologist.
* Subjects will be asked to complete the Dermatology Quality of Life Index (DQLI)
* Use Trichology device to capture images of scalp target area for efficacy assessments
* Collect blood for safety laboratory tests
* Dispense 3-month supply of investigational product
* Provide subjects with instruction for using kit contents
* Remind subjects to follow inclusion/exclusion criteria for restrictions for both OTC and prescription medications, maintain current dietary habits, sleep habits, exercise and sexual intercourse habits
* Provide subjects with a diary to record product use and any changes to health status or medication use
* Subjects will be booked for their next appointment

Visit 5 (Return for anagen/telogen ratio assessment) - day 87 Subjects will return to the clinic to have the anagen/telogen ratio assessed.

Visit 6 - Day 168 Study subjects will return to the Clinic on Day 168.

The following procedures will be completed:

* Collect daily diaries and review
* Collected investigational product containers (used and unused) and assess compliance
* Monitor adverse events (since the previous visit)
* Review concomitant medications (including changes to medications, changes to dose and frequency)
* Measure anthropometrics and vital signs: weight (kg), temperature (°C) respiratory rate (breaths/min), blood pressure (mmHg) and heart rate (bpm)
* Calculate BMI (kg/m2)
* Scalp examination (including photographs) for each subject will include a screen for observable medical issues and any skin/scalp disorders; photography of hair (top, right side, left side, back) - photographs will be reviewed and SALT score determined by a dermatologist.
* Subjects will be asked to complete the Dermatology Quality of Life Index (DQLI)
* Use Trichology device to capture images of scalp target area for efficacy assessments
* Collect blood for safety laboratory tests

Visit 7 (Return for anagen/telogen ratio assessment and end of study assessment) - day 171 Subjects will return to the clinic on day 3 to have the baseline anagen/telogen ratio assessed.

Early Termination/Discontinuation Visit

Subjects may elect to independently withdraw from participation in the study at any time. At a termination visit, subjects will be encouraged to undergo the procedures specified in the final study visit. Reasons for early termination/ discontinuation may include the subject developing any condition which contravenes the original criteria, or, at the discretion of the Principal Investigator (PI), the subject is considered to be unsuitable to continue the study. Individual subjects may have administration temporarily interrupted at the discretion of the PI, e.g. for AEs that are subsequently resolved. Subjects MUST have permanent discontinuation in the following situations:

* The subject had a Grade 3 (severe) or an investigational product-related SAE as determined by the PI
* Subject withdraws consent or refuses further assessment during the study
* Participation in another clinical trial
* Subject lost to follow-up
* Death
* Protocol violation

Unscheduled Visits Any study participant who contacts the investigation site about possible adverse events that are more than minor and/or that persist will be asked to visit the research centre for an assessment as appropriate.

Safety Tests Blood will be collected at V1, V4 and V6 for analysis of safety parameters. Anthropometrics and vital signs are being recorded at study visits number 1, 4, and 6 as measures of safety. Additionally, safety will be assessed by means of reported AEs.

Stopping Rules/Discontinuation The Investigator may withdraw any subject from this research if circumstances arise that warrant doing so. If a subject is withdrawn from the study for any reason, they will be asked to complete an early termination visit.

Permitted/Concomitant Medication(s) Subjects will be questioned about their medication history. The details of any medication taken will be recorded in the case notes and electronic Case Report Form (eCRF). Prescription and over-the-counter (OTC) medications (including supplements) not known to affect study endpoints are permitted.

Thyroid medications will be permitted where dosage has been stable for 6 months prior to the screening visit (V1) and subjects are not expected to have a dosage change during the study period.

Prohibited Medication(s)

Medications that are prohibited include:

* Anabolic steroids in prior 6 months and during the clinical study period
* 5-alpha reductase inhibitors in prior 6 months and during the clinical study period
* Products (including natural health products) and/or devices to promote scalp hair growth (e.g. finasteride, minoxidil, etc.) in 30 days prior to baseline (V2) and during the clinical study period
* Medications that are known to potentially cause hair loss or affect growth as determined by PI in 30 days prior to baseline (V2) and during the clinical study period
* Use of coagulation inhibiting medications (including natural health products) during the clinical study period
* Use of blood pressure lowering medications during the clinical study period
* Use of anti-inflammatory medications, corticosteroids or immunosuppressive drugs taken for more than 2 consecutive weeks in the 3 months prior to baseline (V2) and during the clinical study period

Rescue Medication(s) As this study is investigating the effects of a product in a healthy population, there are no rescue medications in this study.

SELECTION AND WITHDRAWAL OF SUBJECTS NUMBER OF STUDY PARTICIPANTS It is estimated that up to 70 subjects will be screened, in order to identify 46 suitable subjects.

WITHDRAWAL CRITERIA Subjects may withdraw from participation in a study at any time without consequence. If a subject withdraws from the study, the PI will make a reasonable effort to determine the reason for withdrawal from the study, which will be recorded on the eCRF, as will any AEs experienced by the subject.

Personal reasons (Subject-initiated): Participation in the study is optional, and a subject can withdraw from the study at any time, without consequence or prejudice.

Clinical judgment of PI: A subject could also be withdrawn from the study if, in the opinion of the PI, it is not in the subject's best interest to continue (e.g. AEs, need for prohibited medication, illness, etc.). All serious AEs (SAEs) will result in withdrawal from the trial.

Protocol violation: If a subject fails to comply with the protocol they may be removed at the discretion of the PI.

Reasons for withdrawal will be documented as one of the following:

W.1 Subject requests withdrawal from the study. W.2 Subject withdraws consent. W.3 AE makes the continuation of the subject in the study impossible or inadvisable.

W.4 Subject was incorrectly included in the study (discovered after enrollment not to have met the protocol entrance criteria). W.5 Subject is not complying with required study procedures.

ELIGIBILITY:
Inclusion Criteria:

1. Men 18 - 65 years of age at time of screening (V1) (inclusive).
2. Have androgenetic alopecia, diffuse hair loss or self-reported thinning or hair loss for more than 3 months prior to screening (V1).
3. Clinically confirmed to have hair loss or thinning by the investigator via physical exam.
4. In good general health, as determined by the Investigator.
5. Willing and able to attend all study visits.
6. Willing to maintain the same hair style as at the Screening Visit and refrain from chemical treatments on the hair for the duration of the study.
7. Have Fitzpatrick skin type I-IV.
8. Be willing and able to cooperate with the requirements of the study.
9. Willingness to be photographed and provide consent for photographic release.
10. Voluntarily sign and date an informed consent approved by the Institutional Review Board.
11. Be able to complete and understand the various rating instruments in English.
12. Sponsor approved global image assessment of degree of thinning / hair loss.

Exclusion Criteria:

1. Female
2. Clinical diagnosis of scarring forms of alopecia or alopecia areata.
3. Clinical diagnosis on the scalp of psoriasis, scaling, fungal or bacterial infection, lesions, follicular dermatitis, lice, flees or chemical burns, unusual thinning patches, traction alopecia or trichokryptomania, trichothiodystrophy, pili annulati, monilethrix or clear signs of trichodysmorphia, poor nutrition or hygiene.
4. Damage to the skin in or around the assessment areas.
5. Scalp hair loss on the treatment area, due to disease, injury, or medical therapy.
6. History of surgical correction of hair loss on the scalp - hair transplants or hair weave.
7. Are using or have used depilatories, razors, or wax on the scalp to an extent which, in the opinion of the investigator, may interfere with the performance of the study assessments
8. In the opinion of the investigator have very little contrast between hair color and scalp that would make trichometric analyses difficult.
9. Subjects who are planning a family and becoming pregnant with their partners during the course of the study or subjects who are unwilling to use appropriate contraceptives for the duration of the study.
10. Current skin disease or conditions on the treatment area that, in the opinion of the Investigator, might put the subject at risk or interfere with the study conduct or evaluations.
11. Presence of major diseases such as diabetes, endocrine, cardiovascular, renal, or liver disease.
12. History of neurological disease (e.g. Parkinson's disease, stroke, traumatic brain injury, etc.).
13. History of blood clotting disorders or current use of coagulation-inhibiting medications including natural health products (e.g. warfarin, St. John's wort).
14. Hypertension defined as a seated resting systolic blood pressure ≥140 mmHg and/or diastolic blood pressure ≥90 mmHg or current use of blood pressure lowering medications.
15. Recently started (<6 months) using hormone replacement therapy.
16. Use of anabolic steroids or 5-alpha reductase inhibitors in 6 months prior to the baseline visit (V2).
17. Use of any products (prescription, OTC or natural health products) or devices reported and used to promote scalp hair growth (e.g., finasteride or minoxidil, L-Tyrosine) within 90 days prior to the Baseline Visit (V2).
18. Use of any medications (including natural health products) that are known to potentially cause hair loss or affect hair growth within 30 days prior to the Baseline Visit (V2), as determined by PI.
19. History of malignancy (in past 5 years) or undergoing chemotherapy or radiation treatments.
20. A known history of autoimmune disease (e.g. HIV/AIDS, systemic lupus erythematosus, inflammatory bowel disease, alopecia areata, alopecia totalis, etc.), uncontrolled thyroid disease [hyperthyroidism, hypothyroidism; controlled will be permitted if no changes in dosage are required in the 6 months prior to screening (V1)], hepatitis C, or any other disorders that in the opinion of the investigator may interfere with the study treatment.
21. Concurrent or within 3 months of baseline (V2) use of anti- inflammatory medication, corticosteroids, or immunosuppressive drugs taken for more than 2 consecutive weeks
22. Active psychiatric disease (hospitalized within the past 12 months of Screening).
23. Evidence of hepatic or renal dysfunction as evidenced by ALT or aspartate aminotransferase (AST) being ≥ 2 times the upper limit of normal or serum creatinine value ≥ 1.5X the upper limit of normal or other clinically significant abnormal clinical laboratory value, such that patient would be classified as stage 3b or greater of chronic kidney failure (eGFR below 60 ml/mjn/1.73 cm2, albumin-creatinine ratio(ACR) > 3.0 mg/mmol), under treatment for uncontrolled hypertension(HT) and other factors per PI discretion.
24. History of drug or alcohol abuse in the past 12 months prior to Screening.
25. Currently consuming more than 2 standard alcoholic beverages a day. A standard alcoholic beverage is defined as 12 ounces of beer, five (5) ounces of wine, or 1.5 ounces of liquor.
26. Have a known sensitivity or allergy to any ingredients in the test products or placebo products.
27. Any condition or abnormality that, in the opinion of the investigator, would compromise the safety of the subject or the quality of the study data.
28. Participating in or has participated in another research study within 30 days prior to screening with any investigational medical product or natural health product

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2018-04-11 (Actual); Primary Completion 2018-10-23 (Actual); Study Completion 2018-10-23 (Actual)

PRIMARY OUTCOMES:
Change in terminal hair density from baseline to Week 24. | 24 Weeks
  The primary outcome will determine if the increase in terminal hair count per square centimeter from baseline to Week 24 in subjects on ALRV5XR therapy is superior to placebo, at a significance level of 5% (one tail). A two-sample t test will be used to compare differences in the mean increase in terminal hair count from baseline to Week 24 between study arms.
The percentage change in the terminal hair regrowth from baseline to Week 24. | 24 Weeks
  The primary outcome will determine if the percentage change in terminal hair count from baseline to Week 24 in subjects on ALRV5XR therapy is superior to placebo, at a significance level of 5% (one tail). A two-sample t test will be used to compare differences in the mean percentage increase in total terminal hair count from baseline to Week 24 between study arms.

SECONDARY OUTCOMES:
Change in terminal hair density from baseline | Week 12
  The increase in terminal hair count per square centimeter from baseline to Week 24 in subjects on ALRV5XR therapy is superior to placebo, at a significance level of 5% (one tail). A two-sample t test will be used to compare differences in the mean increase in terminal hair count from baseline to Week 12 between study arms.
The percentage change in the terminal hair regrowth from baseline to Week 12. | Week 12
  The percentage change in terminal hair count
Change from baseline in hair width. | Week 12 and 24
  Change from baseline in hair width, as measured by macrophotography [Time Frame: Week 12 and 24
Proportion of subjects achieving a ≥25% increase in hair number count | Week 12 and 24
  Proportion of subjects achieving a ≥25% increase in hair number count from baseline in the area being examined, as measured by macrophotography
Proportion of subjects achieving a ≥50% increase in hair number count | Week 12 and 24
  Proportion of subjects achieving a ≥50% increase in hair number count from baseline in the area being examined, as measured by macrophotography
Proportion of subjects achieving a ≥75% increase in hair number count | Week 12 and 24
  Proportion of subjects achieving a ≥75% increase in hair number count from baseline in the area being examined, as measured by macrophotography
Proportion of subjects achieving a ≥25% increase in Severity of Alopecia Tool (SALT) scores | Week 12 and 24
  Proportion of subjects achieving a ≥25% increase in Severity of Alopecia Tool (SALT) scores from baseline. (SALT scores measure scalp hair loss for terminal hair only: 0: no hair loss; 1: 1-24% hair loss; 2: 25-49% hair loss; 3: 50-74% hair loss; 4: 75-99% hair loss, (4A: 75-90% hair loss, 4B: 91-99% hair loss); 5: 100% hair loss.)
Proportion of subjects achieving a ≥50% increase in Severity of Alopecia Tool (SALT) scores | Week 12 and 24
  Proportion of subjects achieving a ≥50% increase in Severity of Alopecia Tool (SALT) scores from baseline. (SALT scores measure scalp hair loss for terminal hair only: 0: no hair loss; 1: 1-24% hair loss; 2: 25-49% hair loss; 3: 50-74% hair loss; 4: 75-99% hair loss, (4A: 75-90% hair loss, 4B: 91-99% hair loss); 5: 100% hair loss.)
Proportion of subjects achieving a ≥75% increase in Severity of Alopecia Tool (SALT) scores | Week 12 and 24
  Proportion of subjects achieving a ≥75% increase in Severity of Alopecia Tool (SALT) scores from baseline. (SALT scores measure scalp hair loss for terminal hair only: 0: no hair loss; 1: 1-24% hair loss; 2: 25-49% hair loss; 3: 50-74% hair loss; 4: 75-99% hair loss, (4A: 75-90% hair loss, 4B: 91-99% hair loss); 5: 100% hair loss.)
Change in anagen/telogen ratio | Week 12 and 24
  Change in anagen/telogen ratio from baseline to weeks 12 and 24
Dermatology Life Quality Index (DLQI) score | Week 12 and 24
  Dermatology Life Quality Index (DLQI) score. (0, no regrowth; 1, <25% of regrowth; 2, 25%-49% of regrowth; 3, 50%-74% of regrowth; 4, 75%-99% of re- growth; 5, 100% of regrowth)
Proportion of subjects achieving a DLQI patient global assessment score of 3 or above | Week 12 and 24
  Proportion of subjects achieving a DLQI patient global assessment score of 3 or above at week 24 (0, no regrowth; 1, <25% of regrowth; 2, 25%-49% of regrowth; 3, 50%-74% of regrowth; 4, 75%-99% of re- growth; 5, 100% of regrowth)

OTHER OUTCOMES:
To evaluate Safety and Tolerability of ALRV5XR | 24 Weeks
  To compare the rate of non-severe and severe adverse events in subjects treated with the ALRV5XR regimen versus placebo treatment

CONTACTS AND LOCATIONS:
Overall Officials: Luciano Marra (Medical Director), PhD, Study Director — Arbor Life Labs
Locations (1):
- Biometrix, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: Yes
Data to support outcomes
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: After publication
Access Criteria: Contact Sponsor

REFERENCES:
- [Derived] Feldman PR, Fiebig KM, Piwko C, Mints BM, Brown D, Cahan DJ, Guevara-Aguirre J. Safety and efficacy of ALRV5XR in men with androgenetic alopecia: A randomised, double-blinded, placebo-controlled clinical trial. EClinicalMedicine. 2021 Sep 11;40:101124. doi: 10.1016/j.eclinm.2021.101124. eCollection 2021 Oct. PMID 34541479